CLINICAL TRIAL: NCT03454256
Title: Effects of Virtual Reality Rehabilitation in Patients With Total Knee Replacement
Brief Title: Virtual Reality Rehabilitation in Patients With Total Knee Replacement
Acronym: VRRS_KNEE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS San Raffaele Roma (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RP 15/16
Record Dates: First submitted 2018-02-26; First posted 2018-03-05 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: Knee Arthropathy; Total Knee Replacement
Keywords: Virtual Reality; Total Knee Replacement; Proprioception; Balance; Gait

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Reality Group (VRG) (Experimental): The Virtual Reality Group (VRG) will perform the rehabilitation trough the Virtual Reality Rehabilitation system (VRRS, Khymeia,Italy). The patient standing upright on a balance board will practice exercises of vertical position control with a visual biofeedback received from the VRRS and interacting with the serious video-games. The difficulty level of the exercises will increase gradually session by session. Every session will last 45 minutes with a frequency of at least 5 times a week.
  Interventions: Device: Virtual Reality
- Control Group (CG) (No Intervention): The Control Group (CG) will perform the traditional treatment consisting of the exercises of rehabilitation of gait and postural passages, exercises for postural control, and proprioceptive exercises in a vertical position according to the method chosen by the physiotherapist. Every session will last 45 minutes with a frequency of at least 5 times a week.

INTERVENTIONS:
Device: Virtual Reality — Virtual Reality Rehabilitation System
  Other Names: VRRS EVO, Khymeia s.r.l., Italy
  Arms: Virtual Reality Group (VRG)

SUMMARY:
Impaired proprioceptive accuracy could be a risk factor for progression of gait limitations in knee osteoarthritis patients, even after the Total Knee Replacement (TKR). Recent studies on Virtual Reality (VR) in rehabilitation show its efficacy in restoring proprioceptive capacity, postural control and gait. However, literature lacks such studies in TKR patients. This preliminary study aims to evaluate the efficacy of a VR system for the enhancement of motor skills in TKR patients compared to a traditional approach of rehabilitation.

DETAILED DESCRIPTION:
In this randomized controlled trial (RCT), the randomization of the sample will be performed by a local software and in a single blind design. Forty patients will be enrolled and after giving the informed consent, assigned to two groups :

* the experimental group (VRG), which will be undergone to treatment with virtual reality for the recovery of load distribution and proper gait pattern;
* the control group (CG), which will be undergone to a traditional rehabilitation addressed to recovery of correct gait pattern for the same time period as VRG.

Both treatments consist in 15 sessions, at least 5 per week , each lasting 45 minutes. Both VRG or CG will last for 21 days from the start of treatment.

All patients, in adjunction to Virtual Reality Rehabilitation (EG) or Traditional Rehabilitation (CG), will execute a global rehabilitation project, consisting in Physiotherapy, Physical Therapies for pain and inflammation control, and Occupational Therapy, personalized by a multidisciplinary rehabilitation team for a minimum of 150-180 minutes per day, and according to their clinical conditions for them.

The purposes of this study in detail are:

1. Observing differences in the distribution of the bi-podalic load in the group that performs a re-education with virtual reality compared to those who perform the traditional treatment.
2. Observing differences in the recovery time of a correct pattern of gait in the group that performs a re-education with virtual reality compared to those who perform a traditional treatment.
3. Observing changes in neurophysiological patterns in the two groups.

ELIGIBILITY:
Inclusion Criteria:

* recruitment and initial assessment within 10 days of surgery;
* monolateral knee arthroplasty in election;
* collaborating patients who are able to perform the proposed exercise;
* good cardiovascular compensation;
* cognitively intact;
* able to provide informed consent;

Exclusion Criteria:

* no severe cognitive / behavioral deficit;
* refusal or inability to provide informed consent;
* presence of sever cardiorespiratory co-morbidities;
* peripheral and /or central neurological deficits;
* visual deficits;
* presence of serious osteo-arthro-muscular diseases at controlateral lower limb against the prosthetic side;
* complication at surgical wound

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2016-11-08 (Actual); Primary Completion 2019-10-08 (Actual); Study Completion 2019-11-13 (Actual)

PRIMARY OUTCOMES:
Change in Time Up and Go (TUG) | Session 1 (baseline) and session 15 (day 21)
  The TUG is a timed test used to assess mobility, balance, and walking in people with balance impairments. The subject must stand up from a chair (which should not be leaned up against a wall), walk a distance of 3 meters, turn around, walk back to the chair and sit down - all performed as quickly and as safely as possible.

SECONDARY OUTCOMES:
Change in 10 Meter Walk Test (10-MWT) | Session 1 (baseline) and session 15 (day 21)
  The 10-MWT examine the patient's gait speed. Patients will be directed to walk at their preferred maximum but safe speed. Patients will be positioned 1 meter before the start line and instructed to walk the entire distance and past the end line approximately 1 meter. The distance before and after the course are meant to minimize the effect of acceleration and deceleration. Time will be recorded using a stopwatch and recorded to the one hundredth of a second (ex: 2.15 second). The test will be recorded 3 times, with adequate rest in between. The average of the 3 times should be recorded.
Change in Medical Research Council scale (MRC) | Session 1 (baseline) and session 15 (day 21)
  The MRC will be used to evaluate the muscle strength of Quadriceps Femoris (QF) and Tibialis Anterior (TA). The muscle scale grades muscle power on a scale of 0 to 5 in relation to the maximum expected for that muscle.
Change in Visual Analog Scale (VAS) | Session 1 (baseline) and session 15 (day 21)
  VAS is a 0-10 rating scale for pain which is used to gain a subjective report of the intensity of a person's pain. Zero represents "no pain" and ten represents "the most intense pain imaginable". A meaningful change would be plus or minus 3 points.
Change in Barthel Index (BI) | Session 1 (baseline) and session 15 (day 21)
  The BI is an ordinal scale used to measure performance in activities of daily living (ADL). Each performance item is rated on this scale with a given number of points assigned to each level or ranking. It uses ten variables describing ADL and mobility. A higher number is associated with a greater likelihood of being able to live at home with a degree of independence following discharge from hospital.
MiniMental State evaluation (MMSE) | Session 1 (baseline)
  The MMSE (Folstein et al., 1975), is a 30-point questionnaire that is used extensively in clinical and research settings to measure intellectual efficiency disorder as well as cognitive impairment.

OTHER OUTCOMES:
Gait Analysis | Session 1 (baseline) and session 15 (day 21)
  Kinematic and kinetic gait parameters will be calculated from data acquired with a motion capture system (SMART-DX; BTSBioengneering, Italy).
Postural Analysis | Session 1 (baseline) and session 15 (day 21)
  Posturographic parameters will be obtained from the analysis of the center of pressure (COP) trajectories measured by force platforms during standing in both open and closed eyes conditions.

CONTACTS AND LOCATIONS:
Overall Officials: Marco Franceschini, MD, Study Chair — IRCCS Sanraffaele Pisana
Locations (1):
- IRCCS San Raffaele Pisana, Roma, RM, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Knoop J, Steultjens MP, van der Leeden M, van der Esch M, Thorstensson CA, Roorda LD, Lems WF, Dekker J. Proprioception in knee osteoarthritis: a narrative review. Osteoarthritis Cartilage. 2011 Apr;19(4):381-8. doi: 10.1016/j.joca.2011.01.003. Epub 2011 Jan 18. PMID 21251988
- [Background] Laver K, George S, Thomas S, Deutsch JE, Crotty M. Cochrane review: virtual reality for stroke rehabilitation. Eur J Phys Rehabil Med. 2012 Sep;48(3):523-30. Epub 2012 Jun 20. PMID 22713539
- [Background] Fung V, Ho A, Shaffer J, Chung E, Gomez M. Use of Nintendo Wii Fit in the rehabilitation of outpatients following total knee replacement: a preliminary randomised controlled trial. Physiotherapy. 2012 Sep;98(3):183-8. doi: 10.1016/j.physio.2012.04.001. Epub 2012 Jul 10. PMID 22898573
- [Background] Lee M, Suh D, Son J, Kim J, Eun SD, Yoon B. Patient perspectives on virtual reality-based rehabilitation after knee surgery: Importance of level of difficulty. J Rehabil Res Dev. 2016;53(2):239-52. doi: 10.1682/JRRD.2014.07.0164. PMID 27149529
- [Background] Negus JJ, Cawthorne DP, Chen JS, Scholes CJ, Parker DA, March LM. Patient outcomes using Wii-enhanced rehabilitation after total knee replacement - the TKR-POWER study. Contemp Clin Trials. 2015 Jan;40:47-53. doi: 10.1016/j.cct.2014.11.007. Epub 2014 Nov 12. PMID 25460343
- [Background] Levinger P, Zeina D, Teshome AK, Skinner E, Begg R, Abbott JH. A real time biofeedback using Kinect and Wii to improve gait for post-total knee replacement rehabilitation: a case study report. Disabil Rehabil Assist Technol. 2016;11(3):251-62. doi: 10.3109/17483107.2015.1080767. Epub 2015 Sep 4. PMID 26336875
- [Background] Dieppe P, Basler HD, Chard J, Croft P, Dixon J, Hurley M, Lohmander S, Raspe H. Knee replacement surgery for osteoarthritis: effectiveness, practice variations, indications and possible determinants of utilization. Rheumatology (Oxford). 1999 Jan;38(1):73-83. doi: 10.1093/rheumatology/38.1.73. No abstract available. PMID 10334686
- [Background] Koralewicz LM, Engh GA. Comparison of proprioception in arthritic and age-matched normal knees. J Bone Joint Surg Am. 2000 Nov;82(11):1582-8. doi: 10.2106/00004623-200011000-00011. PMID 11097448
- [Derived] Pournajaf S, Goffredo M, Pellicciari L, Piscitelli D, Criscuolo S, Le Pera D, Damiani C, Franceschini M. Effect of balance training using virtual reality-based serious games in individuals with total knee replacement: A randomized controlled trial. Ann Phys Rehabil Med. 2022 Nov;65(6):101609. doi: 10.1016/j.rehab.2021.101609. Epub 2022 Sep 29. PMID 34839056